CLINICAL TRIAL: NCT04360694
Title: RandomizEd ClinicAL triaL on the Efficacy and saFety of Incremental Hemodialysis
Brief Title: RandomizEd ClinicAL triaL on the Efficacy and saFety of Incremental Hemodialysis (REAL-LIFE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: European Renal Association - European Dialysis and Transplant Association (Other)
Responsible Party: Principal Investigator, Loreto Gesualdo, MD, Full Professor of Nephrology University of Bari Aldo Moro - Head of the Nephrology, Dialysis and Transplantation Unit, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REAL LIFE
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: End Stage Renal Disease on Dialysis

STUDY DESIGN:
Intervention Model Description: REAL LIFE is a pragmatic, prospective, multicentre, open label RCT, investigator-initiated, comparing the intervention arm (incremental HD) with the control arm (standard 3HD/wk). It consists in starting the HD treatment adopting the new incremental approach guided by the VTM. The investigators recommend to start and keep on with once-weekly HD, which should be possible until residual renal urea clearance (KRU) falls below 2.5 - 3.0 mL/min/35 L, i.e., glomerular filtration rate (GFR) ≈ 4 mL/min/1.73 m2. Then, HD sessions will be increased to twice-weekly. When KRU falls bellow 1.5 ml/min/35L, dialysis schedule will change to thrice-weekly, as per criteria for progression. It is controlled through usual clinical practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incremental hemodialysis (Experimental): Procedure: Incremental hemodialysis. It consists in reducing the frequency or number of sessions per week with which patients start the HD treatment. The experimental group will start with one session/week, then the number of weekly sessions will be increased to two and later to three as per criteria for progression
  Interventions: Procedure: Incremental hemodialysis
- Conventional hemodialysis (Active Comparator): Procedure: Conventional hemodialysis. It is controlled through usual clinical practice, based on starting the HD treatment with three sessions per week (control group).
  Interventions: Procedure: Conventional hemodialysis

INTERVENTIONS:
Procedure: Incremental hemodialysis — 95 patients will start renal replacement therapy (RRT) with an incremental hemodialysis (once-weekly or twice-weekly) regimen.
  Arms: Incremental hemodialysis
Procedure: Conventional hemodialysis — 95 patients will start renal replacement therapy (RRT) with the standard (thrice-weekly) hemodialysis regimen.
  Arms: Conventional hemodialysis

SUMMARY:
Background: The thrice-weekly hemodialysis (HD) regimen is widely accepted as a standard prescription. The concept of incremental dialysis has been established as a possible alternative for patients with preserved diuresis and end-stage renal failure in need of HD. The main problems related to prescription of incremental HD are an arbitrary use of infrequent regimens and the lack of clear standards for incorporating residual kidney function (RKF) in the assessment of HD dose. Several models have been proposed for prescription of incremental dialysis. The latest, the variable target model (VTM), gives more clinical weight to the RKF and allows less frequent HD treatments at lower RKF. Despite increasing evidence derived from observational studies to support the use of incremental HD, RCTs are lacking and, therefore, urgently needed.

Methods/Design:

The Department of Nephrology, Dialysis and Transplantation of the Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Italy and the EUDIAL Working Group of the European Renal Association - European Dialysis Transplant Association (ERA-EDTA) are starting a randomized clinical trial (RCT) in incident HD patients, whose name is "REAL LIFE", by using the acronym of its whole definition: RandomizEd clinicAL triaL on the effIcacy and saFety of incremental haEmodialysis. REAL LIFE is a pragmatic, prospective, multicentre, open label RCT, investigator-initiated, comparing the intervention arm (incremental HD) with the control arm (standard 3HD/wk). The trial, originally conceived by experts at the Division of Nephrology of the Miulli General Hospital, Acquaviva delle Fonti, Italy, consists in starting the HD treatment adopting the new incremental approach guided by the VTM. The primary outcome is the survival of kidney function, with the event defined as urinary output (UO) ≤ 200 mL/day, confirmed by a further collection after 2 weeks to exclude temporary illness.

Discussion: REAL LIFE will enable the investigators to know with the highest level of scientific evidence the safety and efficacy of an incremental approach to the start of HD treatment.

DETAILED DESCRIPTION:
The majority of dialysis patients starting hemodialysis (HD) are currently treated with a fixed dose thrice-weekly HD (3HD/wk). The 3HD/wk regimen has been assumed, until recently, almost as a dogma in the dialysis community. Incremental HD is based on the simple idea of adjusting its dose according to the metrics of RKF. REAL LIFE is a pragmatic, prospective, multicentre, open label RCT, investigator-initiated, comparing the intervention arm (incremental HD) with the control arm (standard 3HD/wk). A Variable Target Model (VTM) has been suggested, which gives more clinical weight to the RKF and allows less frequent HD treatments in patients with lower RKF. The investigators recommend to start and keep on with once-weekly HD, which should be possible until residual renal urea clearance (KRU) falls below 2.5 - 3.0 mL/min/35 L, i.e., glomerular filtration rate (GFR) ≈ 4 mL/min/1.73 m2.

The primary outcome is the survival of kidney function, with the event defined as urinary output (UO) ≤ 200 mL/day, confirmed by a further collection after 2 weeks to exclude temporary illness. Secondary outcomes are: composite primary cardiovascular endpoint (cardiovascular death, non fatal myocardial infarction and/or or non fatal stroke); intima-media thickness of the carotid arteries; specific cardiomyopathy control; RKF preservation; patients survival; hospital admissions; anemia control; mineral and bone disorder control, and middle molecules removal.

The sample size calculation is based on the primary outcome "presence of anuria". The assumptions for calculating the sample size, derived from data of Teruel Briones et al., are the following:

* Percentage of subjects who developed anuria in the experimental group (incremental HD): 25%
* Percentage of subjects who developed anuria in the control group (standard 3HD/wk): 51%
* Power: 0.8
* Ratio: 1:1
* Non-compliance: 20%
* Total expected sample size: 190 (95 participants in each group)

The assessment of the key kinetic parameters as well as the guide to the selection of operative parameters, as required to get the required equilibrated Kt/V (eKt/V = 1.05), will be done by using SPEEDY, a spreadsheet prescription tool that uses essentially the same equations used by Solute Solver, the software based on the double pool UKM recommended by the 2015 KDOQI guidelines. SPEEDY is freely available at the European Nephrology Portal (ENP).

The link is https://enp-era-edta.org/174/page/home. The control arm includes patients put on a thrice-weekly HD schedule, as detailed above. The dialysis dose (eKt/V) should be about 1.05.

PICO question:

Participants with CKD-EPI GFR ≤ 10 ml/min and daily urine output > 600 ml Intervention: one or two weekly hemodialysis (as detailed above) Comparator: three weekly hemodialysis (as per standard practice and as detailed above) Outcome: Residual renal function

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 18 years
* Start of maintenance hemodialysis treatment due to advanced CKD stage 5D
* Patients who are about to start HD or have already started HD within a period of ≤ 2 weeks
* Glomerular filtration rate <= 10 mL/min/1.73 m2, as estimated by means of CKD-EPI formula.

Exclusion Criteria:

* Age < 18 years
* Acute kidney injury or acute on chronic kidney injury
* eGFR higher than 10 mL/min/1.73 m2
* UO < 600 mL/day
* Already treated with other replacement therapies (peritoneal dialysis or kidney transplant)
* Unable or unwilling to give informed consent.
* Unable to comply with trial procedures, e.g., collection of UO.
* Likely survival prognosis or planned modality or centre transfer < 6 months.
* Patients who are in the waiting list for a living kidney transplant
* Associated diseases: active neoplastic disease; refractory congestive heart failure (type IV NYHA, ejection fraction ≤ 30%) requiring high ultrafiltration volumes per session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants whose kidney function remains >200 ml | 24 months
  The survival of kidney function is defined as a time to the event (anuria): the anuria is defined as urinary output (UO) ≤ 200 mL/day, confirmed by a further collection after 2 weeks to exclude temporary illness

SECONDARY OUTCOMES:
Number of participants who develop cardiovascular death, non fatal myocardial infarction and/or or non fatal stroke (composite outcome) | 24 months
  Cardiovascular death, non fatal myocardial infarction and/or or non fatal stroke
Mean value of intima-media thickness of the carotid arteries of participants at end of treatment and change from beginning to end of treatment | 12 and 24 months
  Echographic evaluation of intima-media thickness of the carotid arteries
Value of left ventricular ejection fraction established with cardiac ultrasound at end of treatment and change from beginning to end of treatment | 12 and 24 months
  Ecocardiography reporting data on the left ventricular ejection fraction (LVEF)
Value of residual kidney function (RKF) preservation established by the slope of decline of residual renal urea clearance | 24 months
  The rate of decline in RKF defined as the slope of decline of residual renal urea clearance
Number of people who die | 24 months
  The follow-up time will be determined in days. It will be defined as the difference in days from the date of the end of the follow-up minus the date of the baseline visit. Events will be counted either as deaths (follow-up of less than 24 months) or as end of the follow-up
Number of people who are hospitalized | 24 months
  The number of admissions will be registered.
Value of hemoglobin in participants at end of treatment and change from beginning to end of treatment | Every month
  The hemoglobin levels (in g/dl) will be measured.
Value of serum phosphorus, calcium and parathyroid hormone in participants at end of treatment and change from beginning to end of treatment | Every month and three months
  Serum phosphorus and calcium levels (in mg/dl), and intact PTH (in pg/dl) will be measured.
Value of serum beta 2 microglobulin (middle molecule) at end of treatment and change from beginning to end of treatment | Every three months
  The rate of change in serum beta 2 microglobulin in time will be evaluated
Value of p-cresyl sulfate and inoxyl sulfate at end of treatment and change from beginning to end of treatment (uraemic toxins variation) | Every six months
  Variation of uremic toxins including p-cresyl sulfate and inoxyl sulfate

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari, Italy

REFERENCES:
- [Result] Casino FG, Basile C. The variable target model: a paradigm shift in the incremental haemodialysis prescription. Nephrol Dial Transplant. 2017 Jan 1;32(1):182-190. doi: 10.1093/ndt/gfw339. PMID 27742823
- [Result] Basile C, Casino FG, Kalantar-Zadeh K. Is incremental hemodialysis ready to return on the scene? From empiricism to kinetic modelling. J Nephrol. 2017 Aug;30(4):521-529. doi: 10.1007/s40620-017-0391-0. Epub 2017 Mar 23. PMID 28337715
- [Result] Basile C, Casino FG; EUDIAL Working Group of ERA-EDTA. Incremental haemodialysis and residual kidney function: more and more observations but no trials. Nephrol Dial Transplant. 2019 Nov 1;34(11):1806-1811. doi: 10.1093/ndt/gfz035. No abstract available. PMID 30805639
- [Result] Casino FG, Basile C. A user-friendly tool for incremental haemodialysis prescription. Nephrol Dial Transplant. 2018 Jun 1;33(6):1074-1075. doi: 10.1093/ndt/gfy081. No abstract available. PMID 29672745
- [Result] Casino FG, Lopez T. The equivalent renal urea clearance: a new parameter to assess dialysis dose. Nephrol Dial Transplant. 1996 Aug;11(8):1574-81. PMID 8856214
- [Result] Teruel-Briones JL, Fernandez-Lucas M, Rivera-Gorrin M, Ruiz-Roso G, Diaz-Dominguez M, Rodriguez-Mendiola N, Quereda-Rodriguez-Navarro C. Progression of residual renal function with an increase in dialysis: haemodialysis versus peritoneal dialysis. Nefrologia. 2013;33(5):640-9. doi: 10.3265/Nefrologia.pre2013.May.12038. English, Spanish. PMID 24089155

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT04360694/Prot_SAP_000.pdf